CLINICAL TRIAL: NCT02349334
Title: CONtrol of Faecal Incontinence Using Distal NeuromodulaTion (CONFIDeNT)
Brief Title: UK Trial of Percutaneous Tibial Nerve Stimulation in Patients With Faecal Incontinence
Acronym: CONFIDeNT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 34825; 09/104/16 (Other Grant/Funding Number: NIHR Health Technology Assessment Programme)
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Faecal Incontinence; Bowel Incontinence
MeSH Terms: conditions — Encopresis; Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham electrical stimulation (Sham Comparator): Sham electrical stimulation to forefoot by TENS
  Interventions: Device: Percutaneous Tibial Nerve Stimulation
- Percutaneous tibial nerve stimulation (Active Comparator): Active PTNS via Urgent PC Neuromodulation device, Uroplasty
  Interventions: Device: Percutaneous Tibial Nerve Stimulation

INTERVENTIONS:
Device: Percutaneous Tibial Nerve Stimulation

SUMMARY:
Faecal incontinence occurs when a person passes faeces (stools) without the usual control. It is a distressing condition that is actually very common although under-reported because of embarrassment. Milder symptoms may be managed by treatments such as dietary change, drugs and bowel retraining, but many patients still resort to surgery to improve symptoms. Although several operations exist to treat incontinence e.g. those aiming to repair damaged anal sphincter muscles, it is now clear that these often have poor results.

Two relatively new treatments called sacral nerve stimulation (SNS) and percutaneous tibial nerve stimulation (PTNS) involve sending pulses of electricity to the nerves controlling the bowel and muscles of the anus (anal sphincter).

SNS does this by inserting electrodes in the lower back just above the tailbone and connecting them to an implanted electrical stimulator which is buried in the buttock and acts a bit like a heart pacemaker. SNS is a relatively well-established treatment in specialist centres, which has been used for over 10 years. It has been shown in studies to be successful for faecal incontinence achieving some improvement in at least three quarters of patients. In Europe, this procedure is fast becoming first treatment offered when non-surgical treatments fail. Nevertheless, SNS is not a miracle cure for all, requiring 2 operations, with potential complications and expensive equipment (> £10,000 approx).

PTNS is a newer treatment, which involves electrically stimulating a nerve at the ankle, using a very small needle, as an outpatient (a bit like acupuncture). This sends signals back to the spine region to try and improve symptoms of faecal incontinence. Since this is a newer treatment, fewer studies have been performed to quantify how successful it is, but early results of PTNS suggest that it may be as good as SNS. If this is true, this is very important because it is much less invasive and considerably cheaper than SNS (equipment £500 per patient).

This project will for the first time determine how effective PTNS is in the treatment of patients with faecal incontinence, by comparing it to sham (fake stimulation). This study is a properly designed clinical trial of 212 patients in at least 14 UK Specialist Centres.. The results of this trial will lead to direct benefits for patients and the NHS.

ELIGIBILITY:
Inclusion Criteria:

* Faecal incontinence sufficiently severe enough to warrant intervention
* Failure of appropriate conservative therapies
* Age ≥ 18 years

Exclusion Criteria:

* Inability to provide informed consent for the research study
* Inability to fill in the detailed bowel diaries required for outcome assessments (this will exclude participants who do not speak / read English)*
* Neurological diseases, such as diabetic neuropathy, multiple sclerosis and Parkinson's disease (any participant with painful peripheral neuropathy)
* Anatomical limitations that would prevent successful placement of needle electrode
* Other medical conditions precluding stimulation: e.g. bleeding disorders, certain cardiac pacemakers, peripheral vascular disease or ulcer, lower leg cellulitis
* Congenital anorectal anomalies or absence of native rectum due to surgery
* A cloacal defect
* Present evidence of external full thickness rectal prolapse
* Previous rectal surgery (rectopexy / resection) done < 12 months ago (24 months for cancer),
* Stoma in situ
* Chronic bowel diseases such as inflammatory bowel disease leading to chronic uncontrolled diarrhoea
* Pregnancy or intention to become pregnant
* Previous experience of SNS or PTNS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome: Binary - success or failure based on % patients achieving > or = 50% reduction in faecal incontinence episodes | 3 months
  From 2 weekly bowel diaries before and after treatment

SECONDARY OUTCOMES:
Reduction in faecal incontinence episodes | 3 months
Proportion of patients achieving >25%, >75% and 100% reduction in faecal incotinence episodes | 3 months
Reduction in Cleveland Clinic Constipation Score | 3 months